CLINICAL TRIAL: NCT04225156
Title: A Phase 3, Multicenter, Open-label, Long-term Trial to Evaluate the Safety and Efficacy of Efgartigimod (ARGX 113) 10 mg/kg Intravenous in Adult Patients With Primary Immune Thrombocytopenia.
Brief Title: A Long-term Study to Assess the Safety and Efficacy of Efgartigimod in Adult Patients With Primary Immune Thrombocytopenia (ITP).
Acronym: ADVANCE+
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-1803; 2019-002101-21 (EudraCT Number)
Record Dates: First submitted 2020-01-06; First posted 2020-01-13 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Primary Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — efgartigimod alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- efgartigimod (Experimental): patients receiving efgartigimod
  Interventions: Biological: efgartigimod

INTERVENTIONS:
Biological: efgartigimod — Intravenous infusion of efgartigimod
  Other Names: ARGX-113

SUMMARY:
This is an open-label long-term multicenter phase 3 trial to evaluate the efficacy and safety of ARGX-113 in adult patients with primary ITP.

ELIGIBILITY:
Inclusion criteria:

1. Ability to understand the requirements of the trial, to provide written informed consent (including consent for the use and disclosure of research-related health information), and to comply with the trial protocol procedures (including required trial visits).
2. Patients enrolled in the ARGX-113-1801 trial who completed the 24-weeks trial period.
3. Women of childbearing potential must have a negative urine pregnancy test at baseline before trial medication (infusion) can be administered.
4. Women of childbearing potential should use a highly effective or acceptable method of contraception during the trial and for 90 days after the last administration of the IMP. They must be on a stable regimen, for at least 1 month (as listed in the protocol)

6. Ability to understand the requirements of the additional 52-week treatment period of the trial, to provide written informed consent (including consent for the use and disclosure of research-related health information), and to comply with the trial protocol procedures (including required trial visits).

7. Patient has completed a 52-week treatment period.

Exclusion criteria:

1. Introduction or continuation of non-permitted medications during the ARGX-113-1801 trial (such as anti-CD20 therapy, romiplostim, monoclonal antibodies, Fc fusion proteins or live/live-attenuated vaccines).
2. Pregnant or lactating women, and those intending to become pregnant during the trial or within 90 days after the last dosing.
3. Patients with known medical history of hypersensitivity to any of the ingredients of efgartigimod.
4. Use of any other investigational drug or participation in any other investigational trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2026-03-11 (Estimated); Study Completion 2026-03-11 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of Adverse Events | Up to 60 weeks
Frequency and severity of vital signs | Up to 60 weeks
Frequency and severity of laboratory assessments | Up to 60 weeks

SECONDARY OUTCOMES:
Extent of disease control defined as the percentage of weeks in the trial with platelet counts of ≥50×10E9/L. | Over the 52 weeks of treatment
Percentage of patients with overall platelet count response defined as achieving a platelet count of ≥50×10^9/L on at least 4 occasions at any time during the 52-week treatment period. | Over the 52 weeks of treatment
Mean change from baseline in platelet count at each visit. | Up to 60 weeks, at each visit
For patients rolling-over from the ARGX-113-1801 trial with a platelet count of <30×10^9/L: time to response is defined as the time to achieve 2 consecutive platelet counts of ≥50×10^9/L | Up to 60 weeks, at each visit
The percentage of weeks in the trial with platelet counts of ≥30×109/L and at least 20×10E9/L above baseline. | Over the 52 weeks of treatment
In patients with baseline platelet count of <15×10E9/L in the current trial (ARGX-113-1803), the percentage of weeks in the trial with platelet counts of ≥30×10E9/L and at least 20×10E9/L above baseline. | Over the 52 weeks of treatment
In patients with first exposure to efgartigimod: proportion of patients who achieve a sustained platelet response defined as achieving platelet counts of at least 50×10^9/L for at least 4 of the 6 visits between week 19 and 24 of the trial. | Up to 5 weeks, between visit 19 and 24 of the trial
In patients with first exposure to efgartigimod: proportion of patients in the overall population achieving platelet counts of at least 50x10^9/L for at least 6 of the 8 visits between week 17 and 24 of the trial. | Up to 7 weeks, between visit 17 and 24 of the trial
Rate of receipt of rescue therapy (rescue per patient per month). | Up to 60 weeks, at each visit
Reduction in concurrent ITP therapy. | Up to 60 weeks, at each visit
Incidence and severity of the WHO-classified bleeding events. | Up to 60 weeks, at each visit
Change from baseline in Patient reported Outcomes (FACIT-Fatigue) at planned visits. | Up to 52 weeks
Change from baseline in Patient reported Outcomes (Fact-Th6) at planned visits. | Up to 52 weeks
Change from baseline in Quality of Life (SF-36) at planned visits. | Up to 52 weeks
Incidence of anti-drug antibodies (ADA) to efgartigimod. | Up to 216 weeks
Pharmacokinetic parameter of efgartigimod: serum concentration observed predose (Ctrough). | Up to 60 weeks
Pharmacodynamics markers: total IgG. | Up to 60 weeks

CONTACTS AND LOCATIONS:
Locations (87):
- United States (4):
  - Investigator Site 0010045, Washington D.C., District of Columbia
  - Investigator Site 0010037, Ocala, Florida
  - Investigator Site 0010042, Iowa City, Iowa
  - Investigator Site 0010040, Columbus, Ohio
- Austria (2):
  - Investigator Site 0430002, Vienna
  - Investigator Site 0430003, Vienna
- Belgium (4):
  - Investigator Site 0320012, Brasschaat
  - Investigator Site 0320011, Bruges
  - Investigator Site 0320014, Turnhout
  - Investigator Site 0320002, Yvoir
- Bulgaria (2):
  - Investigator Site 3590001, Pleven
  - Investigator Site 3590002, Sofia
- Czechia (4):
  - Investigator Site 4200001, Brno
  - Investigator Site 4200008, Olomouc
  - Investigator Site 4200006, Ostrava
  - Investigator Site 4200007, Prague
- France (4):
  - Investigator Site 0330009, Créteil
  - Investigator Site 0330018, Montpellier
  - Investigator Site 0330008, Pessac
  - Investigator Site 0330016, Périgueux
- Georgia (5):
  - Investigator site 9950007, Tbilisi
  - Investigator site 9950008, Tbilisi
  - Investigator site 9950009, Tbilisi
  - Investigator site 9950011, Tbilisi
  - Investigator site 9950012, Tbilisi
- Germany (2):
  - Investigator Site 0490010, Düsseldorf
  - Investigator Site 0490008, Essen
- Hungary (5):
  - Investigator Site 0360004, Budapest
  - Investigator Site 0360006, Debrecen
  - Investigator Site 0360015, Győr
  - Investigator Site 0360010, Nyíregyháza
  - Investigator Site 0360014, Szombathely
- Italy (9):
  - Investigator Site 0390014, Milan
  - Investigator Site 0390020, Monza
  - Investigator Site 0390015, Novara
  - Investigator Site 0390010, Ravenna
  - Investigator Site 0390011, Reggio Calabria
  - Investigator Site 0390018, Reggio Emilia
  - Investigator Site 0390019, Rimini
  - Investigator Site 0390009, Siena
  - Investigator Site 0390016, Trieste
- Japan (9):
  - Investigator Site 0810015, Hirakata
  - Investigator Site 0810010, Hiroshima
  - Investigator Site 0810017, Iruma
  - Investigator Site 0810022, Kashiwa
  - Investigator Site 0810018, Maebashi
  - Investigator Site 0810021, Niigata
  - Investigator Site 0810014, Sapporo
  - Investigator Site 0810016, Shibukawa
  - Investigator Site 0810023, Shimotsuke
- Netherlands (2):
  - Investigator Site 0310005, Rotterdam
  - Investigator Site 0310006, The Hague
- Poland (5):
  - Investigator Site 0480012, Gdansk
  - Investigator Site 0480013, Katowice
  - Investigator Site 0480011, Lodz
  - Investigator Site 0480014, Lublin
  - Investigator Site 0480026, Nowy Sącz
- Russia (7):
  - Investigator Site 0070006, Kaluga
  - Investigator Site 0070008, Moscow
  - Investigator Site 0070007, Petrozavodsk
  - Investigator Site 0070013, Rostov-on-Don
  - Investigator Site 0070015, Syktyvkar
  - Investigator Site 0070012, Tula
  - Investigator Site 0070010, Ufa
- Spain (9):
  - Investigator Site 0340006, Barcelona
  - Investigator Site 0340007, Barcelona
  - Investigator Site 0340009, Madrid
  - Investigator Site 0340014, Madrid
  - Investigator Site 0340012, Palma de Mallorca
  - Investigator Site 0340015, Pozuelo de Alarcón
  - Investigator Site 0340013, Seville
  - Investigator Site 0340004, Valencia
  - Investigator Site 0340011, Valencia
- Turkey (Türkiye) (11):
  - Investigator Site 0900003, Ankara
  - Investigator Site 0900006, Ankara
  - Investigator Site 0900015, Ankara
  - Investigator Site 0900016, Edirne
  - Investigator Site 0900013, Istanbul
  - Investigator Site 0900004, Izmir
  - Investigator Site 0900010, Mersin
  - Investigator Site 0900007, Sakarya
  - Investigator Site 0900009, Samsun
  - Investigator Site 0900017, Tekirdağ
  - Investigator Site 0900019, Trabzon
- Investigator Site 3800006, Mykolaiv, Ukraine
- United Kingdom (2):
  - Investigator Site 0440008, London
  - Investigator Site 0440012, Southampton

IPD SHARING:
Plan to Share IPD: Undecided